CLINICAL TRIAL: NCT06560216
Title: Effects of Supplementation of Cryopreservation Medium With Apigenin on Post-thaw Human Sperm
Brief Title: Cryopreservation Medium With Apigenin on Post-thaw Human Sperm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 062267
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Apigenin; Cryopreservation; Antioxidant; Human sperm; Oxidative stress
MeSH Terms: interventions — Apigenin

STUDY DESIGN:
Intervention Model Description: 1. Frozen-thawed control without apigenin supplementation in freezing medium
  2. Frozen-thawed sperm suspension with apigenin supplementation in freezing medium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Frozen-thawed sperm suspension without apigenin supplementation in freezing medium
- Apigenin (Experimental): Frozen-thawed sperm suspension with apigenin 0.2 mM supplementation in freezing medium
  Interventions: Dietary Supplement: Apigenin

INTERVENTIONS:
Dietary Supplement: Apigenin — 0.2 mM in freezing medium
  Arms: Apigenin

SUMMARY:
The goal of this clinical trial is to compare the effect of apigenin supplementation in freezing medium with no apigenin supplementation in freezing medium on post-thaw human sperm motility. It will also evaluate the sperm viability, total antioxidant capacity, and oxidative stress markers. The main questions it aims to answer are:

* Does apigenin supplementation in freezing medium improve the post-thaw sperm motility?
* Does apigenin supplementation in freezing medium improve the post-thaw sperm viability, total antioxidant capacity, and oxidative stress?

DETAILED DESCRIPTION:
All normal semen samples from participants who give written informed consent and meet the eligibility requirements will be included in the study. Prepared semen samples were divided into 3 groups.

1. Pre-freezing sperm suspension
2. Frozen-thawed control without apigenin supplementation in freezing medium
3. Frozen-thawed sperm suspension with apigenin 0.2 mM supplementation in freezing medium Baseline sperm motility will be measured in pre-freezing sperm suspension. The last 2 groups will be stored in liquid nitrogen for at least one week. After thawing, the sperm suspensions will be evaluated for motility, viability, total antioxidant capacity, and oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-45 years who can receive semen analysis services at the Reproductive Biology Unit, Chulalongkorn Hospital, Thai Red Cross Society
* Normal semen analysis results according to the World Health Organization criteria (Volume ≥ 1.4 mL, Sperm concentration ≥ 16 million/mL, Total motility ≥ 42%, Progressive motility ≥ 30%)
* Giving consent

Exclusion Criteria:

* A history of accidents, radiation to the testes, or a history of male reproductive system surgery
* Undescended testis
* Varicocele
* A history of taking certain medications that affect sperm production, such as chemotherapy, hormones
* Currently having sexually transmitted disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Percentage of sperm motility | At least 1 week of freezing
  Sperm motility (total motility, progressive motility, non-progressive motility, immotile spermatozoa) will be reported in percentage.
  Compare results among freezing medium with apigenin group, control group, and baseline pre-freeze sperm suspension.

SECONDARY OUTCOMES:
Percentage of sperm viability comparison between intervention and control group | At least 1 week of freezing
  Viability test will be assessed by eosin-nigrosin staining technique

OTHER OUTCOMES:
Total antioxidant capacity comparison between intervention and control group | At least 1 week of freezing
  Total antioxidant capacity will be assessed by ABTS assay
Oxidative stress markers comparison between intervention and control group | At least 1 week of freezing
  Oxidative stress markers will be measured. e.g. reactive oxygen species

CONTACTS AND LOCATIONS:
Overall Officials: Punyawee Utaipatanacheep, Principal Investigator — Chulalongkorn University
Locations (2):
- Thailand (2):
  - Chulalongkorn Hospital, Bangkok
  - Chulalongkorn University, Bangkok

IPD SHARING:
Plan to Share IPD: No
You can ask for information directly from the investigators.

REFERENCES:
- [Background] PubChem [Internet]. Bethesda (MD): National Library of Medicine (US), National Center for Biotechnology Information; 2004-. PubChem Compound Summary for CID 5280443, Apigenin; [cited 2024 July 25]. [Internet]. 2004. Available from: https://pubchem.ncbi.nlm.nih.gov/compound/Apigenin.
- [Background] World Health Organization. WHO laboratory manual for the examination and processing of human semen. 6th ed. Geneva: World Health Organization, Cop; 2021.
- [Background] Ngamjarus C, Pattanittum P. n4Studies: application for sample size calculation in health science research. Version 2.3. App store. 2024.
- [Background] Ngamjarus C. Sample size calculation for health science research. 1st ed. Khon Kaen University Printing House, Khon Kaen, Thailand 2021.
- [Background] Chow S-C, Shao J, Wang H. Sample size calculations in clinical research. 2 ed. Boca Raton: FLA: Chapman and Hall/CRC; 2003.
- [Result] Anger JT, Gilbert BR, Goldstein M. Cryopreservation of sperm: indications, methods and results. J Urol. 2003 Oct;170(4 Pt 1):1079-84. doi: 10.1097/01.ju.0000084820.98430.b8. PMID 14501696
- [Result] Sharma Y, Sharma M. Sperm Cryopreservation: Principles and Biology. J Infertil Reprod Biol 2020;8:43-8.
- [Result] Hai E, Li B, Zhang J, Zhang J. Sperm freezing damage: the role of regulated cell death. Cell Death Discov. 2024 May 18;10(1):239. doi: 10.1038/s41420-024-02013-3. PMID 38762505
- [Result] Keel BA, Black JB. Reduced motility longevity in thawed human spermatozoa. Arch Androl. 1980 May;4(3):213-5. doi: 10.3109/01485018008986965. PMID 7416844
- [Result] O'Connell M, McClure N, Lewis SE. The effects of cryopreservation on sperm morphology, motility and mitochondrial function. Hum Reprod. 2002 Mar;17(3):704-9. doi: 10.1093/humrep/17.3.704. PMID 11870124
- [Result] Ozkavukcu S, Erdemli E, Isik A, Oztuna D, Karahuseyinoglu S. Effects of cryopreservation on sperm parameters and ultrastructural morphology of human spermatozoa. J Assist Reprod Genet. 2008 Aug;25(8):403-11. doi: 10.1007/s10815-008-9232-3. Epub 2008 Aug 13. PMID 18704674
- [Result] Oberoi B, Kumar S, Talwar P. Study of human sperm motility post cryopreservation. Med J Armed Forces India. 2014 Oct;70(4):349-53. doi: 10.1016/j.mjafi.2014.09.006. Epub 2014 Oct 16. PMID 25382909
- [Result] Liu T, Gao J, Zhou N, Mo M, Wang X, Zhang X, Yang H, Chen Q, Ao L, Liu J, Cui Z, Cao J. The effect of two cryopreservation methods on human sperm DNA damage. Cryobiology. 2016 Jun;72(3):210-5. doi: 10.1016/j.cryobiol.2016.04.004. Epub 2016 Apr 25. PMID 27126062
- [Result] Hezavehei M, Sharafi M, Kouchesfahani HM, Henkel R, Agarwal A, Esmaeili V, Shahverdi A. Sperm cryopreservation: A review on current molecular cryobiology and advanced approaches. Reprod Biomed Online. 2018 Sep;37(3):327-339. doi: 10.1016/j.rbmo.2018.05.012. Epub 2018 Aug 22. PMID 30143329
- [Result] Darsini N, Hamidah B, Suyono S, Ashari F, Aswin R, Yudiwati R. Human Sperm Motility, Viability, and Morphology Decreased after Cryopreservation. Folia Medica Indonesiana 2019;55:198.
- [Result] Fernandez-Lopez P, Garriga J, Casas I, Yeste M, Bartumeus F. Predicting fertility from sperm motility landscapes. Commun Biol. 2022 Sep 28;5(1):1027. doi: 10.1038/s42003-022-03954-0. PMID 36171267
- [Result] Wang S, Wang W, Xu Y, Tang M, Fang J, Sun H, Sun Y, Gu M, Liu Z, Zhang Z, Lin F, Wu T, Song N, Wang Z, Zhang W, Yin C. Proteomic characteristics of human sperm cryopreservation. Proteomics. 2014 Feb;14(2-3):298-310. doi: 10.1002/pmic.201300225. PMID 24259508
- [Result] Amidi F, Pazhohan A, Shabani Nashtaei M, Khodarahmian M, Nekoonam S. The role of antioxidants in sperm freezing: a review. Cell Tissue Bank. 2016 Dec;17(4):745-756. doi: 10.1007/s10561-016-9566-5. Epub 2016 Jun 24. PMID 27342905
- [Result] Agarwal A, Rana M, Qiu E, AlBunni H, Bui AD, Henkel R. Role of oxidative stress, infection and inflammation in male infertility. Andrologia. 2018 Dec;50(11):e13126. doi: 10.1111/and.13126. PMID 30569652
- [Result] Sudhakaran G, Kesavan D, Kandaswamy K, Guru A, Arockiaraj J. Unravelling the epigenetic impact: Oxidative stress and its role in male infertility-associated sperm dysfunction. Reprod Toxicol. 2024 Mar;124:108531. doi: 10.1016/j.reprotox.2023.108531. Epub 2024 Jan 2. PMID 38176575
- [Result] Antioxidants in Sperm Cryopreservation , bookTitle= Male Infertility: Contemporary Clinical Approaches, Andrology, ART and Antioxidants. Cham: Springer International Publishing; 2020. 671--8 p.
- [Result] Sabeti P, Pourmasumi S, Rahiminia T, Akyash F, Talebi AR. Etiologies of sperm oxidative stress. Int J Reprod Biomed. 2016 Apr;14(4):231-40. PMID 27351024
- [Result] Mannucci A, Argento FR, Fini E, Coccia ME, Taddei N, Becatti M, Fiorillo C. The Impact of Oxidative Stress in Male Infertility. Front Mol Biosci. 2022 Jan 5;8:799294. doi: 10.3389/fmolb.2021.799294. eCollection 2021. PMID 35071326
- [Result] Barranco I, Tvarijonaviciute A, Perez-Patino C, Parrilla I, Ceron JJ, Martinez EA, Rodriguez-Martinez H, Roca J. High total antioxidant capacity of the porcine seminal plasma (SP-TAC) relates to sperm survival and fertility. Sci Rep. 2015 Dec 21;5:18538. doi: 10.1038/srep18538. PMID 26688188
- [Result] Di Santo M, Tarozzi N, Nadalini M, Borini A. Human Sperm Cryopreservation: Update on Techniques, Effect on DNA Integrity, and Implications for ART. Adv Urol. 2012;2012:854837. doi: 10.1155/2012/854837. Epub 2011 Dec 13. PMID 22194740
- [Result] Moubasher AE, El Din AM, Ali ME, El-sherif WT, Gaber HD. Catalase improves motility, vitality and DNA integrity of cryopreserved human spermatozoa. Andrologia. 2013 Apr;45(2):135-9. doi: 10.1111/j.1439-0272.2012.01310.x. Epub 2012 May 16. PMID 22591546
- [Result] Tas DO, Ozkavukcu S, Inanc I, Kose SK, Erdemli E. The effects of coenzyme Q10 and curcumin supplementation in freezing medium for human sperm cryopreservation. Eur J Obstet Gynecol Reprod Biol. 2023 Aug;287:36-45. doi: 10.1016/j.ejogrb.2023.05.040. Epub 2023 Jun 2. PMID 37276727
- [Result] Moradi Gardeshi T, Shahandeh E, Tavakolpoor Saleh N, Karami S, Mirzaei Azandaryani Z, Mazaheri F, Mohammadi H. Evaluation of the effect of mitoquinone on functional parameters, DNA structure, and genes expression related to the apoptotic and antioxidants of human sperm after freezing-thawing. Mol Biol Rep. 2024 Jan 23;51(1):183. doi: 10.1007/s11033-023-09020-0. PMID 38261086
- [Result] Jannatifar R, Asa E, Sahraei SS, Verdi A, Piroozmanesh H. N-acetyl-l-cysteine and alpha lipoic acid are protective supplement on human sperm parameters in cryopreservation of asthenoteratozoospermia patients. Andrologia. 2022 Dec;54(11):e14612. doi: 10.1111/and.14612. Epub 2022 Nov 1. PMID 36321244
- [Result] Akbarzadeh-Jahromi M, Jafari F, Parsanezhad ME, Alaee S. Evaluation of supplementation of cryopreservation medium with gallic acid as an antioxidant in quality of post-thaw human spermatozoa. Andrologia. 2022 Dec;54(11):e14571. doi: 10.1111/and.14571. Epub 2022 Aug 23. PMID 36054457
- [Result] Noto D, Collodel G, Cerretani D, Signorini C, Gambera L, Menchiari A, Moretti E. Protective Effect of Chlorogenic Acid on Human Sperm: In Vitro Studies and Frozen-Thawed Protocol. Antioxidants (Basel). 2021 May 7;10(5):744. doi: 10.3390/antiox10050744. PMID 34067222
- [Result] Mohammadi F, Varanloo N, Heydari Nasrabadi M, Vatannejad A, Amjadi FS, Javedani Masroor M, Bajelan L, Mehdizadeh M, Aflatoonian R, Zandieh Z. Supplementation of sperm freezing medium with myoinositol improve human sperm parameters and protects it against DNA fragmentation and apoptosis. Cell Tissue Bank. 2019 Mar;20(1):77-86. doi: 10.1007/s10561-018-9731-0. Epub 2019 Jan 29. PMID 30694450
- [Result] Najafi L, Halvaei I, Movahedin M. Canthaxanthin protects human sperm parameters during cryopreservation. Andrologia. 2019 Nov;51(10):e13389. doi: 10.1111/and.13389. Epub 2019 Aug 11. PMID 31402476
- [Result] Aghaz F, Khazaei M, Vaisi-Raygani A, Bakhtiyari M. Cryoprotective effect of sericin supplementation in freezing and thawing media on the outcome of cryopreservation in human sperm. Aging Male. 2020 Dec;23(5):469-476. doi: 10.1080/13685538.2018.1529156. Epub 2018 Nov 19. PMID 30453816
- [Result] Ghorbani M, Amiri I, Khodadadi I, Fattahi A, Atabakhsh M, Tavilani H. Influence of BHT inclusion on post-thaw attributes of human semen. Syst Biol Reprod Med. 2015 Jan;61(1):57-61. doi: 10.3109/19396368.2014.968267. Epub 2014 Oct 6. PMID 25285571
- [Result] Saeednia S, Bahadoran H, Amidi F, Asadi MH, Naji M, Fallahi P, Nejad NA. Nerve growth factor in human semen: Effect of nerve growth factor on the normozoospermic men during cryopreservation process. Iran J Basic Med Sci. 2015 Mar;18(3):292-9. PMID 25945243
- [Result] Li Z, Lin Q, Liu R, Xiao W, Liu W. Protective effects of ascorbate and catalase on human spermatozoa during cryopreservation. J Androl. 2010 Sep-Oct;31(5):437-44. doi: 10.2164/jandrol.109.007849. Epub 2009 Oct 15. PMID 19834132
- [Result] Noegroho BS, Siregar S, Tampubolon KAG. Antioxidant Supplementation on Sperm DNA Fragmentation and Sperm Parameters: A Systematic Review and Meta-Analysis. Turk J Urol. 2022 Sep;48(5):375-384. doi: 10.5152/tud.2022.22058. PMID 36197144
- [Result] Bahmyari R, Zare M, Sharma R, Agarwal A, Halvaei I. The efficacy of antioxidants in sperm parameters and production of reactive oxygen species levels during the freeze-thaw process: A systematic review and meta-analysis. Andrologia. 2020 Apr;52(3):e13514. doi: 10.1111/and.13514. Epub 2020 Jan 21. PMID 31967363
- [Result] Mushtaq Z, Sadeer N, Hussain M, Mahwish, Alsagaby S, Imran M, et al. Therapeutical properties of apigenin: a review on the experimental evidence and basic mechanisms. International Journal of Food Properties 2023;26:1914-39.
- [Result] Bhardwaj H, Vasudeva N, Sharma S. Phytochemistry And Pharmacological Aspects Of Apigenin: A Review. The Natural Products Journal 2022;12.
- [Result] Balez R, Steiner N, Engel M, Munoz SS, Lum JS, Wu Y, Wang D, Vallotton P, Sachdev P, O'Connor M, Sidhu K, Munch G, Ooi L. Neuroprotective effects of apigenin against inflammation, neuronal excitability and apoptosis in an induced pluripotent stem cell model of Alzheimer's disease. Sci Rep. 2016 Aug 12;6:31450. doi: 10.1038/srep31450. PMID 27514990
- [Result] Shukla S, Gupta S. Apigenin: a promising molecule for cancer prevention. Pharm Res. 2010 Jun;27(6):962-78. doi: 10.1007/s11095-010-0089-7. Epub 2010 Mar 20. PMID 20306120
- [Result] Raskovic A, Gigov S, Capo I, Paut Kusturica M, Milijasevic B, Kojic-Damjanov S, Martic N. Antioxidative and Protective Actions of Apigenin in a Paracetamol-Induced Hepatotoxicity Rat Model. Eur J Drug Metab Pharmacokinet. 2017 Oct;42(5):849-856. doi: 10.1007/s13318-017-0407-0. PMID 28255865
- [Result] Nafisi S, Hashemi M, Rajabi M, Tajmir-Riahi HA. DNA adducts with antioxidant flavonoids: morin, apigenin, and naringin. DNA Cell Biol. 2008 Aug;27(8):433-42. doi: 10.1089/dna.2008.0735. PMID 18491957
- [Result] Sharma H, Kanwal R, Bhaskaran N, Gupta S. Plant flavone apigenin binds to nucleic acid bases and reduces oxidative DNA damage in prostate epithelial cells. PLoS One. 2014 Mar 10;9(3):e91588. doi: 10.1371/journal.pone.0091588. eCollection 2014. PMID 24614817
- [Result] Kopalli SR, Yoo SK, Kim B, Kim SK, Koppula S. Apigenin Isolated from Carduus crispus Protects against H2O2-Induced Oxidative Damage and Spermatogenic Expression Changes in GC-2spd Sperm Cells. Molecules. 2022 Mar 8;27(6):1777. doi: 10.3390/molecules27061777. PMID 35335140
- [Result] Dang Y, Li Z, Luo B, Pan L, Wei Q, Zhang Y. Protective effects of apigenin against acrylonitrile-induced subchronic sperm injury in rats. Food Chem Toxicol. 2017 Nov;109(Pt 1):517-525. doi: 10.1016/j.fct.2017.09.025. Epub 2017 Sep 28. PMID 28963002
- [Result] Shi Y, Bai J, Dang Y, Bai Q, Zheng R, Chen J, Li Z. Protection of apigenin against acrylonitrile-induced sperm and testis injury in rats: involvement of activation of ASK1-JNK/p38 signaling pathway. Toxicol Res (Camb). 2021 Mar 11;10(2):159-168. doi: 10.1093/toxres/tfab017. eCollection 2021 Mar. PMID 33884167
- [Result] Pei Y, Yang L, Wu L, He H, Geng G, Xu D, Chen H, Li Q. Combined effect of apigenin and ferulic acid on frozen-thawed boar sperm quality. Anim Sci J. 2018 Jul;89(7):956-965. doi: 10.1111/asj.13009. Epub 2018 Apr 30. PMID 29708294
- [Result] Wang H, Lu P, Yuan C, Zhao J, Liu H, Lu W, Wang J. Effects of Apigenin and Astragalus Polysaccharide on the Cryopreservation of Bull Semen. Animals (Basel). 2021 May 22;11(6):1506. doi: 10.3390/ani11061506. PMID 34067384
- [Result] Mohammadi T, Hosseinchi Gharehaghaj M, Alaei Novin A. Effects of apigenin and trans-ferulic acid on microscopic and oxidative stress parameters in the semen of water buffalo bulls during cryopreservation. Cryobiology. 2024 Jun;115:104868. doi: 10.1016/j.cryobiol.2024.104868. Epub 2024 Feb 27. PMID 38423495
- [Result] Najafi A, Mohammadi H, Sharifi SD, Rahimi A. Apigenin supplementation substantially improves rooster sperm freezability and post-thaw function. Sci Rep. 2024 Feb 24;14(1):4527. doi: 10.1038/s41598-024-55057-x. PMID 38402367
- [Result] Esmaeili Irani A, Nikoozar B, Arbabian M, Tavalaee M, Nasr-Esfahani MHa. The Antioxidant Effect of Apigenin on Human Sperm Quality after Freezing-Thawing. Journal of Gorgan University of Medical Sciences 2024;26.
- [Result] Auger J, Kunstmann JM, Czyglik F, Jouannet P. Decline in semen quality among fertile men in Paris during the past 20 years. N Engl J Med. 1995 Feb 2;332(5):281-5. doi: 10.1056/NEJM199502023320501. PMID 7816062
- [Result] Aribarg A, Sukcharoen N, Chanprasit Y, Ngeamvijawat J. Prediction of post-thaw sperm motility and sperm cryosurvival rate using the pre-freeze sperm parameters. J Med Assoc Thai. 1995 Sep;78(9):474-80. PMID 7561575